CLINICAL TRIAL: NCT04445688
Title: Phase 2, Randomized, 3-Period, Placebo-Controlled Crossover Study to Evaluate the Efficacy and Safety in Obstructive Sleep Apnea of AD036 Versus Placebo or Atomoxetine
Brief Title: Crossover Trial of AD036 in Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APN-006
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AD036 (Experimental): AD036 oral capsule administered before sleep
  Interventions: Drug: AD036
- Atomoxetine (Active Comparator): Atomoxetine oral capsule administered before sleep
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Placebo oral capsule administered before sleep
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AD036 — Oral administration before bed
  Arms: AD036
Drug: Atomoxetine — Oral administration before bed
  Arms: Atomoxetine
Drug: Placebo — Oral administration before bed
  Arms: Placebo

SUMMARY:
This is a randomized, 3-Period, Placebo-Controlled, Crossover, phase 2 clinical study to examine the efficacy and safety of AD036 versus placebo or atomoxetine in patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
The study is designed to examine the efficacy and safety of AD036 to treat obstructive sleep apnea. The study is a three-period single-dose randomized crossover design in which patients will undergo overnight Home Sleep Apnea Testing (HSAT) with dosing of one of the following 3 treatments: AD036, Atomoxetine, or Placebo. Participants will return 1 week after their final crossover HSAT for an end of study (EOS) Visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, between 25 to 65 years of age, inclusive, at the Screening Visit.
* AHI 10 to <20, or AHI ≥20 if meets PSG criteria

Exclusion Criteria:

* History of narcolepsy.
* Clinically significant craniofacial malformation.
* Clinically significant cardiac disease (e.g., rhythm disturbances, coronary artery disease or cardiac failure) or hypertension requiring more than 2 medications for control. A medication for these purposes is defined by dosage form, such that a combination antihypertensive medication is considered 1 medication
* CPAP should not be used for at least 2 weeks prior to first study PSG
* History of using oral or nasal devices for the treatment of OSA may enroll as long as the devices are not used during participation in the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - SDS Clinical Trials, Inc., Santa Ana, California
  - The Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Sleep Medicine & Research Center, St. Luke's Hospital, Chesterfield, Missouri
  - CTI Clinical Research Center, Cincinnati, Ohio

REFERENCES:
- [Result] Schweitzer PK, Maynard JP, Wylie PE, Emsellem HA, Sands SA. Efficacy of atomoxetine plus oxybutynin in the treatment of obstructive sleep apnea with moderate pharyngeal collapsibility. Sleep Breath. 2023 May;27(2):495-503. doi: 10.1007/s11325-022-02634-x. Epub 2022 May 13. PMID 35551600

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 clinical sites screened 101 participants 62 were randomized. This was an unblinded three period placebo controlled study. Participants who withdrew were not replaced.
Pre-assignment Details: All participants were centrally randomized to one of 6 sequences (A - B - C, B - C - A, C - B - A, A - C - B, B - A - C, C - A - B). A 1-week minimum washout period occurred between each of the 3 arm assignments.
Groups:
- All Participants: oral capsules administered before bedtime. Treatment A: AD036, Treatment B: atomoxetine + placebo, Treatment C: placebo + placebo
Period: First Intervention
Arm/Group | All Participants
Started | 62
Treatment A | 21
Treatment B | 21
Treatment C | 20
Completed | 62
Not Completed | 0
Period: Washout (One Week)
Arm/Group | All Participants
Started | 62
Completed | 59
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Period: Second Intervention
Arm/Group | All Participants
Started | 59
Treatment A | 18
Treatment B | 21
Treatment C | 20
Completed | 59
Not Completed | 0
Period: Washout (One Week)
Arm/Group | All Participants
Started | 59
Completed | 59
Not Completed | 0
Period: Third Intervention
Arm/Group | All Participants
Started | 59
Treatment A | 20
Treatment B | 20
Treatment C | 19
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 59
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 53 [28 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 41
  More than one race | 1
  Unknown or Not Reported | 0
BMI (kg/m^2) [Median (Full Range); unit: kg/m^2] | 32.30 [22.6 to 39.6]

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index
Description: Apnea-Hypopnea Index(Disease severity is often defined based on the number of apneas and hypopneas per hour during sleep), AD036 vs. placebo
Time Frame: 1 day
Population: The efficacy was analyzed using the mITT Population comprised of all participants who took at least 1 dose of any of the study treatments and had at least 1 measurement on the primary endpoint. Sixty (96.8%) patients were included in the mITT Population. Patients were analyzed for efficacy according to the treatment sequence into which they were randomized. Due to insufficient data quality of the home sleep test, AHI could not be determined in some treatment conditions.
Measure: Least Squares Mean (95% Confidence Interval); unit: events/hour
Arm/Group | AD036 | Atomoxetine | Placebo
Number analyzed (Participants) | 54 | 56 | 57
events/hour | 11.5 [7.2 to 15.8] | 11.5 [7.2 to 15.8] | 18.8 [14.5 to 23.1]
Statistical Analysis 1: Comparison: AD036 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; difference in Least Squares Mean = -7.3, 95% CI 2-sided [-10.2 to -4.4]

2. Secondary Outcome: Hypoxic Burden
Description: Hypoxic burden (a way to measure oxygen desaturation) determined by measuring the respiratory event-associated area under the desaturation curve from pre-event baseline, AD036 vs. placebo. Hypoxic Burden was measured during polysomnography (type of sleep study), while the patient was asleep
Time Frame: 1 day
Population: The efficacy was analyzed using the mITT Population comprised of all participants who took at least 1 dose of any of the study treatments and had at least 1 measurement on the primary endpoint. Sixty (96.8%) patients were included in the mITT Population. Patients were analyzed for efficacy according to the treatment sequence into which they were randomized. Due to insufficient data quality of the home sleep test, hypoxic burden could not be determined in some treatment conditions.
Measure: Least Squares Mean (95% Confidence Interval); unit: %min/hour
Arm/Group | AD036 | Atomoxetine | Placebo
Number analyzed (Participants) | 54 | 56 | 57
%min/hour | 24.3 [13.5 to 35.1] | 26.8 [16.1 to 37.6] | 46.1 [35.4 to 56.8]
Statistical Analysis 1: Comparison: AD036 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; difference in Least Squares Mean = -21.8, 95% CI 2-sided [-29.5 to -14.1]

3. Secondary Outcome: ODI
Description: Oxygen Desaturation Index, measured by pulse-oximetry, AD036 vs. placebo
Time Frame: 1 day
Population: The efficacy was analyzed using the mITT Population comprised of all participants who took at least 1 dose of any of the study treatments and had at least 1 measurement on the primary endpoint. Sixty (96.8%) patients were included in the mITT Population. Patients were analyzed for efficacy according to the treatment sequence into which they were randomized. Mean (SD) of ODI (4%). Due to insufficient data quality of the home sleep test, ODI could not be determined in some treatment conditions.
Measure: Least Squares Mean (95% Confidence Interval); unit: events/hour
Arm/Group | AD036 | Atomoxetine | Placebo
Number analyzed (Participants) | 54 | 56 | 57
events/hour | 12.8 [8.4 to 17.1] | 13.3 [9.0 to 17.7] | 20.1 [15.8 to 24.4]
Statistical Analysis 1: Comparison: AD036 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; difference in Least Squares Mean = -7.3, 95% CI 2-sided [-10.5 to -4.2]

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Planned time points for all adverse events assessments at each study visit
Arm/Group | AD036 | Atomoxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/62 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/62 | 0/59
Other Adverse Events (participants affected / at risk) | 8/59 | 11/62 | 5/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AD036 (N=59) | Atomoxetine (N=62) | Placebo (N=59)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT04445688/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT04445688/SAP_001.pdf